CLINICAL TRIAL: NCT02400645
Title: Comparison of Laparoscopically Assisted Transversus Abdominis Plane Block Using Liposomal Bupivacaine With Pre-incisional Bupivacaine for Post-operative Pain Control in Patients Undergoing Laparoscopic or Robotic Hysterectomy
Brief Title: TAP Block With Liposomal Bupivacaine Versus Pre-incisional Wound Infiltration With Bupivacaine for Postoperative Pain
Acronym: LATAP
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: It was determined that one member of the team had falsified data.
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-132
Record Dates: First submitted 2015-03-11; First posted 2015-03-27 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2015-03

CONDITIONS: Postoperative Pain
Keywords: laparoscopic hysterectomy; robotic assisted hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: pre-incisional bupivacaine (Active Comparator): Intervention: Pre-incisional wound infiltration with bupivacaine plain 0.25%. Ketorolac 30mg IV will be given following surgical procedure.
  Interventions: Procedure: Pre-incisional wound infiltration; Drug: Bupivacaine; Drug: Ketorolac
- Group B: laparoscope to place TAP block (Active Comparator): Intervention: laparoscope to place TAP block with liposomal bupivacaine and bupivacaine plain 0.25%. Ketorolac 30 mg IV will be given following surgical procedure.
  Interventions: Procedure: Laparoscope to place TAP block with liposomal bupivacaine; Drug: Liposomal bupivacaine; Drug: Bupivacaine; Drug: Ketorolac

INTERVENTIONS:
Procedure: Pre-incisional wound infiltration — Intraoperative: Pre-incisional bupivacaine 0.25% up to 20 cc divided dose for trocar incisions
  Arms: Group A: pre-incisional bupivacaine
Procedure: Laparoscope to place TAP block with liposomal bupivacaine — Intraoperative: Laparoscopic TAP block with Liposomal bupivacaine and bupivacaine 0.25%
  Other Names: Laparoscopic TAP block with Liposomal bupivacaine
  Arms: Group B: laparoscope to place TAP block
Drug: Liposomal bupivacaine — Use of Liposomal bupivacaine in laparoscopic TAP block
  Other Names: Exparel
  Arms: Group B: laparoscope to place TAP block
Drug: Bupivacaine — 20 cc Bupivacaine 0.25% plain will be used for either pre-incisional injection or added to laparoscopic TAP block solution.
  Other Names: Marcaine
Drug: Ketorolac — Ketorolac 30mg to be given IV at end of surgical procedure unless contraindicated.
  Other Names: Toradol

SUMMARY:
In this randomized, controlled, double-blinded trial we plan to evaluate post-operative pain relief after laparoscopic-assisted Transversus Abdominis Plane (TAP) block using liposomal bupivacaine plus bupivacaine versus pre-incisional would infiltration with bupivacaine in patients undergoing Total laparoscopic or robotic assisted laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Patients undergoing laparoscopic or robotic assisted total hysterectomy at Erlanger Hospital will be randomized into one of two groups to receive either laparoscopic assisted TAP block with liposomal bupivacaine and bupivacaine (Group A) or pre-incisional bupivacaine (Group B). The remaining aspects of the perioperative care, including the general anesthesia care and postoperative care will be similar for all patients. Ideally, patients will be informed and consented for the study in the preoperative clinic setting. They will be randomized in the pre-anesthesia care unit.

Patients in Group A will receive laparoscopic-assisted bilateral TAP blocks using 10cc liposomal bupivacaine, 10cc Bupivacaine 0.25% and 10cc Normal Saline one each side. Patients in Group B will receive a total of 20cc pre-incisional Bupivacaine divided between each of the trocar sites. All patients will receive Ketorolac 30 mg, IV at the conclusion of surgery. All patients will be offered either oral pain medications or patient controlled anesthesia (PCA) opiate pain medication as indicated. Morphine equivalents will be calculated.

Postoperative pain control will be assessed using Visual Analog Pain Score (VAS). This will be done by recovery room personnel who will be blinded as to whether the patients received TAP block or pre-incisional anesthetic. VAS will be assessed at rest at 1 hour and 2 hours after arrival to PACU. Patients will be assessed with Overall Benefit of Anesthesia Score (OBAS) questionnaires at postoperative days 1, 2 and 7. OBAS questionnaires will be done by personnel blinded to anesthesia technique. Patients will also be blinded as to which group they were in. Total morphine equivalents of intraoperative and postoperative pain medications will be calculated through postoperative day 7.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3,
* Scheduled for laparoscopic or robotic assisted laparoscopic hysterectomy,
* Able to participate personally or by legal representation in informed consent

Exclusion Criteria:

* History of relevant allergy to the study drugs (Bupivacaine),
* Chronic opioid use or drug abuse history,
* Inability to understand the study protocol,
* Refusal to provide written consent,
* Soft tissue infection of the abdominal wall and skin

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog pain scores (VAS) | Two hours
  1. Postoperative pain at 1 hour and 2 hours after arrival to recovery using Visual Analog Pain Scores (VAS)
  2. VAS: 0 (no pain) TO 10 (worst possible pain)

SECONDARY OUTCOMES:
Narcotic pain medication usage | 2 hours postoperative
  Narcotic pain medication usage intraoperative and in recovery assessed as morphine equivalents
Narcotic pain medication following surgery | 1 week
  Narcotic pain medication pill counts up to one week postoperatively

OTHER OUTCOMES:
Overall Benefit of Anesthesia scores (OBAS) on postoperative days 1,2 and 7 | One week
  1. Overall Benefit of Anesthesia Scores (OBAS) Questionnaires at postoperative days 1,2 and 7.
  2. OBAS covers pain, vomiting, itching, sweating, freezing, dizziness and overall satisfaction on a scale of 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Shanti I Mohling, MD, Principal Investigator — University of Tennessee